CLINICAL TRIAL: NCT06730620
Title: Bioequivalence Study of Methacholine for Inhalation
Brief Title: Bioequivalence Study of Methacholine Chloride
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ting YANG, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TQC3610-BE-01
Record Dates: First submitted 2024-11-30; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Healthy People
MeSH Terms: interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test preparation：Methylcholine chloroacetate for inhalation (Experimental): Inhale methacholine solution for 1 minute
  Interventions: Drug: Test preparation：Methylcholine chloroacetate for inhalation
- Reference preparation：Methylcholine chloroacetate for inhalation（(Provocholin） (Active Comparator): Inhale methacholine solution for 1 minute
  Interventions: Drug: Reference preparation：Methylcholine chloroacetate for inhalation（(Provocholin）

INTERVENTIONS:
Drug: Test preparation：Methylcholine chloroacetate for inhalation — Cholinergic agonists
  Arms: Test preparation：Methylcholine chloroacetate for inhalation
Drug: Reference preparation：Methylcholine chloroacetate for inhalation（(Provocholin） — Cholinergic agonists
  Arms: Reference preparation：Methylcholine chloroacetate for inhalation（(Provocholin）

SUMMARY:
This trial was divided into two parts. The first part was the PK bioequivalence study in healthy people, which was designed as a single-dose, randomized, open, four-cycle, two-sequence, fully repeated crossover design, and planned to enroll 20 subjects.

ELIGIBILITY:
Inclusions Criteria

1. Male or female healthy subjects aged 18 to 50 years old (including 18 and 50 years old).
2. Male subjects weigh no less than 50 kg, female subjects weigh no less than 45 kg; and body mass index (BMI) = weight (kg) / height 2 (m2), and body mass index is within the range of 18.5~27.0 (including critical values).

3) Normal pulmonary function test (FEV1 ≥ 80% predicted value, FEV1/FVC ≥ 0.7), FEV1 decline rate after inhalation of saline is no more than 20%, and methacholine chloride provocation test is negative.

4. Sign the informed consent form before the experiment and fully understand the content, process and possible adverse reactions of the experiment.

5. Subjects can communicate well with researchers and understand and comply with the requirements of this study.

Exclusions Criteria

1. Ask for any diseases that might interfere with the test results
2. Have a history of drug/food allergy
3. blood collection difficulties or can not tolerate indwelling needle blood collection
4. Patients who had surgery within 4 weeks prior to the trial or planned to have surgery during the study period
5. Patients who have used any drug within 2 weeks before the test
6. Subjects have participated in any drug or medical device clinical study within 3 months prior to screening (except those who failed screening or did not receive any experimental drug).
7. Blood loss or blood donation exceeding 400 mL in the 3 months prior to screening (excluding female menstrual blood loss), or who intend to donate blood during the trial or within 1 month after the trial.
8. pregnant and lactating women, or pregnancy test positive.
9. Male subjects (or their partners) or female subjects had unprotected sex or had a pregnancy plan from 1 week before screening to 3 months after the end of the trial, and were unwilling to use one or more non-drug contraceptive methods (such as total abstinence, contraceptive rings, partner ligation, etc.) during the trial.
10. Previous history of drug abuse/drug use; Or test positive for drug abuse.
11. the diet has special requirements, can not comply with the unified diet.
12. Those who had a smoking history within 6 months before the test, smoked more than 5 cigarettes per day, or were unwilling to give up smoking during the test, or had positive results of nicotine screening.
13. Alcoholics or regular drinkers in the six months prior to the trial, i.e. drinking more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or breath-positive for alcohol.
14. Eating a diet within 48 hours prior to taking the study drug that may affect the metabolism of the drug in the body, smoking, drinking behavior, or other diet that the investigator believes may affect the absorption, distribution, metabolism, or excretion of the drug.
15. Physical examination, electrocardiogram, laboratory examination, vital signs and other tests related to the test were judged by the investigator to be abnormal and clinically significant.
16. Acute illness or concomitant medication occurred from the screening stage to the study medication.
17. Subjects who may not be able to complete the study for other reasons or who the investigator believes should not be included

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-02-03 (Actual)

PRIMARY OUTCOMES:
Peak Concentration | Within 60 minutes before administration and within 3 minutes, 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 6 hours, and 8 hours after administration
  The highest plasma drug concentration that can be achieved after administration
The area under the blood concentration time curve when the time is from 0 to the last time point selected（AUC0-t） | Within 60 minutes before administration and within 3 minutes, 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 6 hours, and 8 hours after administration
  The area under the blood concentration time curve from 0 to t after administration
The area under the blood concentration time curve during time from 0 to infinity（AUC0-∞） | Within 60 minutes before administration and within 3 minutes, 5 minutes, 10 minutes, 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 6 hours, and 8 hours after administration
  Area under the blood concentration time curve after medication

CONTACTS AND LOCATIONS:
Locations (1):
- China-japan Friendship Hospital, Beijing, Beijing Municipality, China